CLINICAL TRIAL: NCT04853407
Title: A Phase III, A Multicenter, Double-blind, Randomized, Placebo-controlled Study Verify the Efficacy and Safety of Ansofaxine Hydrochloride Extended-release Tablets for Major Depressive Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Ansofaxine Hydrochloride Extended-release Tablets in the Treatment of Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03005/CT-CHN-305
Record Dates: First submitted 2021-04-08; First posted 2021-04-21 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LY03005 extended-release tablets 80 mg group (Experimental): orally once a day
  Interventions: Drug: LY03005 extended-release tablet
- LY03005 extended-release tablets 160 mg group (Experimental): orally once a day
  Interventions: Drug: LY03005 extended-release tablet
- Placebo group (Placebo Comparator): orally once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY03005 extended-release tablet — orally once a day
  Arms: LY03005 extended-release tablets 160 mg group; LY03005 extended-release tablets 80 mg group
Drug: Placebo — orally once a day
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine if LY03005 is effective and safe in improve MADRS score, as compared to placebo (no medicine) in participants with Major Depressive Disorder (MDD)

DETAILED DESCRIPTION:
The study consisted of two periods: a screening period of 1 week and a double-blind treatment period (8 weeks). After the screening period, 588 enrolled subjects were randomized into one of 3 study groups in the 1:1:1 ratio, 2 LY03005 treatment groups with different dose or 1 placebo group. Subjects were given investigatory drug or placebo according to the protocol, followed up at the end of 1, 2, 4 6, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 65 years subjects from outpatients;
2. Subjects currently meet the Diagnostic and Statistical Manual of Manual Disorders, fifth Edition(DSM-5) criteria for MDD with either single or recurrent episodes (296.2/296.3) without psychotic characteristics;
3. Subjects has a total score of the Montgomery- Åsberg Depression Scale (MADRS) ≥26 points at screening;
4. Subjects has a clinical Global Impression -severity illness (CGI-S) score≥4 points at screening

Exclusion Criteria:

1. Allergic or known to be allergic to venlafaxine and desvenlafaxine;
2. Subjects with MDD who were not responsive to the previous venlafaxine treatment with sufficient amount and duration and to at least two different mechanisms of action antidepressants with adequate amount and duration in the past;
3. There is a clear suicide attempt or behavior and score of the 10th item (suicidal ideation) in MADRS scale is 4 points or greater;
4. Pregnant or lactating women,women who have a planned pregnancy in the near future;
5. Subjects meet the diagnostic criteria for other psychotic disorders(except for MDD) in DSM-5, such as Schizophrenia Spectrum and Other Psychotic Disorders, Bipolar and Related Disorders, Obsessive-Compulsive and related Disorders, post-traumatic stress disorder, separation disorders, anorexia nervosa or bulimia and personality disorder;
6. Subjects who meet the diagnostic criteria for substance or alcohol abuse (excluding nicotine or caffeine) 6 months prior to the screening;
7. MDD secondary to other mental illnesses or physical illnesses;
8. Those with a history of seizures (except for convulsions caused by febrile seizures in children).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Montgomery- Åsberg Depression Rating Scale(MADRS) | 8 Weeks
  Changes from baseline in the 10-items Montgomery- Åsberg Depression Scales (MADRS) total scores at the end of treatment.
  The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).

SECONDARY OUTCOMES:
17 items Hamilton Depression Scales (HAM-D17) | 8 Weeks
  Changes from baseline in the 17 items Hamilton Depression Scales (HAM-D17) total scores at the end of treatment.
  HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Nine items are scored on a 3 point scale (0=none/absent to 2=most severe) and 8 items are scored on a 5 point scale (0=none/absent to 4=most severe) for a maximum total score of 50; higher score indicates more depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Zhang, Principal Investigator — Peking University Sixth Hospital
Locations (1):
- The Sixth Hospital of Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mi W, Di X, Wang Y, Li H, Xu X, Li L, Wang H, Wang G, Zhang K, Tian F, Luo J, Yang C, Zhou Y, Xie S, Zhong H, Wu B, Yang D, Chen Z, Li Y, Chen J, Lv S, Yi Q, Jiang Z, Tian J, Zhang H. A phase 3, multicenter, double-blind, randomized, placebo-controlled clinical trial to verify the efficacy and safety of ansofaxine (LY03005) for major depressive disorder. Transl Psychiatry. 2023 May 10;13(1):163. doi: 10.1038/s41398-023-02435-0. PMID 37164957